CLINICAL TRIAL: NCT04845009
Title: The Effectiveness of Progressive Muscle Relaxation on Postoperative Pain, Fatigue, and Vital Signs in Patients With Head and Neck Cancers
Brief Title: Relaxation Therapy for Pain, Fatigue and Vital Signs in Post-operation With Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: relaxation for HN
Record Dates: First submitted 2021-04-12; First posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Progressive Muscle Relaxation on Postoperative Pain, Fatigue, and Vital Signs in Patients With Head and Neck Cancers
Keywords: progressive muscle relaxation; head and neck cancer
MeSH Terms: conditions — Fatigue; Head and Neck Neoplasms | interventions — Autogenic Training

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- progressive muscle relaxation (Experimental): progressive muscle relaxation tape guided
  Interventions: Behavioral: progressive muscle relaxation
- usual care (Placebo Comparator): usual care
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: progressive muscle relaxation — progressive muscle relaxation
  Arms: progressive muscle relaxation
Behavioral: Usual care — Usual care
  Arms: usual care

SUMMARY:
This study aimed to investigate the effects of progressive muscle relaxation (PMR) on postoperative pain, fatigue, and vital signs in patients with head and neck cancers.

ELIGIBILITY:
Inclusion Criteria:

- Head and neck cancer, need for surgery.

(1) clear consciousness; (2) >= 20 years; (3) no history of surgery for head and neck cancer, regardless of cancer staging, tracheostomy tubing, degree of primary tumor resection, neck dissection, modified radical neck dissection, resection of cervical nerve root branches, and flap reconstruction (including free flap and transposition flap); (4) plan to undergo surgery; (5) willingness to participate in this study and provide informed consent; (6) physically capable of participation the study, as determined by the physician in charge; (7) ability to communicate in Mandarin or Taiwanese, with no reading, listening, or writing disability, and complete the questionnaire alone or with the assistance of the researchers.

Exclusion Criteria:

- Head and neck cancer, not for surgery.

(1) use of hypnotics or record of a sleep disorder within 3 months prior to admission; (2) difficulty hearing, external auditory canal trauma, or hearing impairment; (3) diagnosis of a psychotic disorder or cognitive impairment; (4) experience practicing Jacobson's PMR.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2016-05-20 (Actual); Study Completion 2016-05-20 (Actual)

PRIMARY OUTCOMES:
Pain level change | preoperative day to postoperative day 10
  The VAS (visual analog scale) score of pain levels, range 0-100, higher score means more severe symptoms.
muscle tightness level change | preoperative day to postoperative day 10
  The VAS (visual analog scale) score of muscle tightness levels, range 0-100, higher score means more severe symptoms.
Fatigue levels change | preoperative day to postoperative day 10
  The VAS (visual analog scale) score of fatigue levels, range 0-100, higher score means more severe symptoms.

SECONDARY OUTCOMES:
Heart rate change | preoperative day to postoperative day 10
  Heart rate change
Systolic blood pressure change | preoperative day to postoperative day 10
  Systolic blood pressure change
Diastolic blood pressure change | preoperative day to postoperative day 10
  Diastolic blood pressure change
Anxiety level | preoperative day to postoperative day 10
  The VAS (visual analog scale) score of Anxiety levels, range 0-100, higher score means more severe symptoms.
depression level | preoperative day to postoperative day 10
  The VAS (visual analog scale) score of depression levels, range 0-100, higher score means more severe symptoms.
sleep disturbance level | preoperative day to postoperative day 10
  The VAS (visual analog scale) score of sleep disturbance levels, range 0-100, higher score means more severe symptoms.